CLINICAL TRIAL: NCT05853939
Title: Inducing and Measuring Visual-evoked Potential Plasticity in Humans With Repetitive Transcranial Magnetic Stimulation
Brief Title: Measuring rTMS-induced Neuroplasticity With EEG Steady-state Visual-evoked Potentials
Status: Enrolling by invitation | Phase: Not Applicable | Type: Interventional
Sponsor: Stanford University (Other)
Collaborators: National Eye Institute (NEI) (NIH)
Responsible Party: Principal Investigator, Ryan T. Ash MD, PhD, Instructor, Stanford University
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Basic Science
Other Study IDs: 62922
Record Dates: First submitted 2023-05-02; First posted 2023-05-11 (Actual); Last update posted 2024-04-22 (Actual); Status verified 2024-04

CONDITIONS: Visual Cortical Plasticity; Repetitive Transcranial Magnetic Stimulation; Visual Attention
Keywords: visual-evoked potentials; TMS; neuroplasticity
MeSH Terms: interventions — Transcranial Magnetic Stimulation

STUDY DESIGN:
Intervention Model Description: Cross-over: 1 Hz vs 10 Hz vs sham rTMS; stimulation to attended or unattended hemisphere
Who Masked: Participant
Masking Description: Participant is blind to the rTMS target hemisphere, the rTMS stimulation parameters, and the objective of the study
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes

ARMS (6):
- Visual Cortex, 1 Hz rTMS, Attended (Experimental)
  Interventions: Device: repetitive transcranial magnetic stimulation
- Visual Cortex, 1 Hz rTMS, Unattended (Experimental)
  Interventions: Device: repetitive transcranial magnetic stimulation
- Visual Cortex, 10 Hz rTMS, Attended (Experimental)
  Interventions: Device: repetitive transcranial magnetic stimulation
- Visual Cortex, 10 Hz rTMS, Unattended (Experimental)
  Interventions: Device: repetitive transcranial magnetic stimulation
- Visual Cortex, Sham, Attended (Sham Comparator)
  Interventions: Device: repetitive transcranial magnetic stimulation
- Visual Cortex, Sham, Unattended (Sham Comparator)
  Interventions: Device: repetitive transcranial magnetic stimulation

INTERVENTIONS:
Device: repetitive transcranial magnetic stimulation — Repetitive TMS targeted by neuronavigation to left lower visual field of primary visual cortex. Randomized to 10 Hz or 1 Hz on different treatment days. Stimulation at 110% of phosphene threshold, or 110% resting motor threshold if phosphenes not detectable. 1 Hz: 1000 pulses total over 1000 seconds. 10 Hz: 1000 pulses over 10 10 second pulse trains, with 50 second intertrain intervals

SUMMARY:
The goals of this study are to 1) use EEG steady-state visual evoked potentials as a noninvasive measure of the neuroplasticity induced by repetitive transcranial magnetic stimulation (rTMS), 2) use visual contrast detection paradigms as a behavioral measure of rTMS effects, and 3) to investigate how visual spatial attention augments or suppresses the neuroplastic impact of rTMS. Participants will observe visual stimuli on a screen while allocating their attention to different parts of the visual field and making responses when they observe changes in the visual stimuli. rTMS is performed to visual cortex using MRI-retinotopy neuronavigation. Then the visual task paradigm is performed again.

ELIGIBILITY:
Inclusion Criteria:

* Men and women, ages 18 to 65
* Must comprehend English well to ensure adequate comprehension of the EEG and TMS instructions, and of clinical scales
* Left- or Right-handed
* No current or history of neurological disorders
* No seizure disorder or risk of seizures

Exclusion Criteria:

* Those with a contraindication for MRIs (e.g. implanted metal)

  * Any unstable medical condition
  * History of head trauma with loss of consciousness
  * History of seizures
  * Neurological or uncontrolled medical disease
  * Active substance abuse
  * Diagnosis of psychotic or bipolar disorder
  * Currently taking medications that substantially reduce seizure threshold (e.g., bupropion, olanzapine, chlorpromazine, lithium)
  * Currently pregnant or breastfeeding

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2023-07-01 (Actual); Primary Completion 2027-05 (Estimated); Study Completion 2027-05 (Estimated)

PRIMARY OUTCOMES:
post-rTMS change in ssVEP Response Amplitude | 60 minutes
  Change in ssVEP contrast-response amplitude after rTMS
post-rTMS change in visual contrast perceptual sensitivity | 60 minutes
  change in visual psychometric threshold across contrasts after rTMS

CONTACTS AND LOCATIONS:
Locations (1):
- Stanford University, Stanford, California, United States

IPD SHARING:
Plan to Share IPD: Yes
The results of this research will be made available via publication in scientific journals and through scientific meetings where our findings are reported. Publication of data shall occur during the project, if appropriate, or at the end of the project, consistent with normal scientific practices. All publications will be made publicly available consistent with NIH policies. Research data, which documents, supports and validates research findings, will be made available after the main findings from the final research data set have been accepted for publication.
Supporting Information: Study Protocol, Analytic Code
Time Frame: Data will be available on reasonable request following completion of data collection.
Access Criteria: see above